CLINICAL TRIAL: NCT05100290
Title: Predictive Properties of the Hyperventilation Provocation Test for the Diagnosis of the Hyperventilation Syndrome
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Université Libre de Bruxelles (Other); Hopitaux Iris Sud (Unknown)
Responsible Party: Sponsor
Other Study IDs: B076201836758-1
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Hyperventilation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HVS+: Subjects without documented respiratory or cardiac disease, with a spirometry and metacholine tests within expected values AND with complaints documented by a Nijmegen questionnaire score of ≥23/64 (suspected of idiopathic hyperventilation)
  Interventions: Diagnostic Test: Hyperventilation Provocation Test (HPTest)
- HVS-: Healthy controls without documented respiratory or cardiac disease, with a spirometry and metacholine tests within expected values AND without complaints documented by a Nijmegen questionnaire score of <23/64
  Interventions: Diagnostic Test: Hyperventilation Provocation Test (HPTest)

INTERVENTIONS:
Diagnostic Test: Hyperventilation Provocation Test (HPTest) — During the HPTest, the subject is comfortably seated in a chair with armrests and breathes in a mouthpiece with a salivary collector and a nasal clamp. Parameters of ventilation and gas exchange are analyzed via an Oxycon ProTM (SN808008) with TripleV-Volume Sensor digital(Jaeger).
  The HPTest begins with a 3-minutes adaptation phase during which the patient is asked to "breathe normally". During the 3-minutes of voluntary hyperventilation phase, the patient is asked to increase his tidal volume and support a breath rate of at least 30/min in order to reduce his PETCO2 by at least 50%. During the recovery phase of the HPTest, the patient is invited to regain a "natural breathing" for 5 minutes, without guidance on tidal volume or breath rate.

SUMMARY:
The Hyperventilation Provocation Test (HPTest) associated with end-tidal CO2 pressure (PETCO2) measurement is a diagnostic tool for idiopathic hyperventilation syndrome (HVS). However, interpretation of HPTest remains unclear regarding the relevant PETCO2 values to consider and the occurrence of subjective symptoms.

This case-control study aims to identify accurate HPTest measurements for the diagnosis of HVS, regardless of symptoms occurrence.

DETAILED DESCRIPTION:
In a first stage, the investigators will analyze in a prospective way a training cohort of HPTest datas from 74 subjects, involving 37 subjects with complaints and a Nijmegen questionnaire score of ≥23/64 (HVS+) matched on gender, age, height, weight and BMI category with 37 healthy controls without complaints and a Nijmegen questionnaire score of <23/64 (HVS-)(16).

All data will have to be collected by the same equipment and by the same operators in the pulmonology department of the CHU-St Pierre-Brussels between June 2018 and October 2021.

To rule out confounding respiratory pathology, each participant will have completed spirometry and methacholine testing, that will have a result within expected normal values.

For both cohorts, kinetics of the PETCO2 recorded during each of the 3 phases of the HPTest (adaptation, hyperventilation and recovery) will be mathematically modeled by an curvilinear model with the parameters (A, A', a and a') noted from the kinetic equation (TAU) : TAU [PETCO2(t)〖=A+a(1-exp〗^((b-t)/c))]. For any observed differences in parameters between groups, the Area Under Curves will be estimated at the cut-off that offers the best Sensitivity and Specificity. False negative and false positive rates will be estimated.

The probability of a type I error is set at 5%.

In a second stage, in order to confirm/infirm the results, a retrospective validation cohort from another care setting, including subjects without confounding pathology, who completed a Nijmegen questionnaire and a HVTest between 2018 and 2021, will be analysed in the same way than the training cohort.

ELIGIBILITY:
Inclusion Criteria:

* Anyone over 18 years of age who has completed an HPTest and a Nijmegen questionnaire between 2015 and 2020

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visited the pulmonary department and performed a HPTest on medical prescription
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
PetCO2 recovery (5min) | 5 minute of recovery
  PetCO2 at the end (5th minute) of the recovery phase of the HPTest

SECONDARY OUTCOMES:
PetCO2 recovery (3min) | 3 minute of recovery
  PetCO2 at the end (3d minute) of the recovery phase of the HPTest

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ninane, Study Director — CHU St PIerre
Locations (1):
- CHU St Pierre, Brussels, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided